CLINICAL TRIAL: NCT04834869
Title: COVID-19 Vaccines Safety Tracking: Global Consortium Study
Brief Title: COVID-19 Vaccines Safety Tracking (CoVaST)
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Other Study IDs: CoVaST
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2021-10

CONDITIONS: Adverse Reaction to Vaccine; COVID19 Vaccine
Keywords: COVID-19; Vaccines; Safety; Side Effects
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; ChAdOx1 nCoV-19; sinovac COVID-19 vaccine; Gam-COVID-Vac vaccine; Ad26COVS1; CVnCoV COVID-19 vaccine; NVX-CoV2373 adjuvated lipid nanoparticle; BBV152 COVID-19 vaccine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (11):
- Pfizer-BioNTech COVID-19 Vaccine: Recently vaccinated individuals by Pfizer-BioNTech COVID-19 Vaccine (Comirnaty)
  Interventions: Biological: BNT162b2
- Moderna COVID-19 Vaccine: Recently vaccinated individuals by Moderna COVID-19 Vaccine
  Interventions: Biological: mRNA-1273
- AstraZeneca-Oxford University COVID-19 Vaccine: Recently vaccinated individuals by AstraZeneca-Oxford University COVID-19 Vaccine (Vaxzevria)
  Interventions: Biological: AZD1222
- CoronaVac: Recently vaccinated individuals by CoronaVac (Sinovac COVID-19 Vaccine)
  Interventions: Biological: CoronaVac
- Sinopharm: Recently vaccinated individuals by Vero Cells (Sinopharm COVID-19 Vaccine)
  Interventions: Biological: Sinopharm
- Sputnik V: Recently vaccinated individuals by Sputnik V COVID-19 Vaccine
  Interventions: Biological: Gam-COVID-Vac
- Janssen: Recently vaccinated individuals by Janssen COVID-19 Vaccine
  Interventions: Biological: JNJ-78436735
- CureVac: Recently vaccinated individuals by CureVac COVID-19 Vaccine
  Interventions: Biological: CVnCoV
- Novavax: Recently vaccinated individuals by Novavax COVID-19 Vaccine
  Interventions: Biological: NVX-CoV2373
- Covaxin: Recently vaccinated individuals by Covaxin COVID-19 Vaccine
  Interventions: Biological: BBV152
- CanSino: Recently vaccinated individuals by CanSino COVID-19 Vaccine

INTERVENTIONS:
Biological: BNT162b2 — Receiving either the first dose only or both doses of BNT162b2 vaccine (Pfizer-BioNTech COVID-19 Vaccine)
  Groups: Pfizer-BioNTech COVID-19 Vaccine
Biological: mRNA-1273 — Receiving either the first dose only or both doses of mRNA-1273 vaccine (Moderna COVID-19 Vaccine)
  Groups: Moderna COVID-19 Vaccine
Biological: AZD1222 — Receiving either the first dose only or both doses of AZD1222 vaccine (AstraZeneca-Oxford University COVID-19 Vaccine)
  Groups: AstraZeneca-Oxford University COVID-19 Vaccine
Biological: CoronaVac — Receiving either the first dose only or both doses of CoronaVac (Sinovac COVID-19 Vaccine)
  Groups: CoronaVac
Biological: Sinopharm — Receiving either the first dose only or both doses of Sinopharm Vero Cell COVID-19 Vaccine
  Groups: Sinopharm
Biological: Gam-COVID-Vac — Receiving either the first dose only or both doses of Gam-COVID-Vac (Sputnik V)
  Groups: Sputnik V
Biological: JNJ-78436735 — Receiving JNJ-78436735 (Janssen COVID-19 Vaccine)
  Groups: Janssen
Biological: CVnCoV — Receiving either the first dose only or both doses of CVnCoV (CureVac COVID-19 vaccine)
  Groups: CureVac
Biological: NVX-CoV2373 — Receiving either the first dose only or both doses of NVX-CoV2373 (Novavax COVID-19 vaccine)
  Groups: Novavax
Biological: BBV152 — Receiving either the first dose only or both doses of BBV152 (Covaxin COVID-19 vaccine)
  Groups: Covaxin

SUMMARY:
This project aims to monitor the side effects of COVID-19 vaccines worldwide actively. The primary objectives of the project include a) to estimate the prevalence of each local and systemic side effect of each COVID-19 vaccine among healthcare workers (HCW), old adults over +65 (OA), and schoolteachers (ST); b) to evaluate the potential demographic and medical risk factors for side effects frequency and intensity; c) to evaluate the long-term consequences of COVID-19 vaccines. The secondary objectives include a) to evaluate the relative safety of COVID-19 vaccines compared to each other; b) to evaluate the impact of palliative drugs used by the recently vaccinated individuals on their short-term side effects resolution.

DETAILED DESCRIPTION:
Introduction:

COVID-19 vaccines are the foremost asset to overcome the ongoing pandemic; therefore, mass vaccination has become a high priority for the world's governments. While vaccination strategies need to be accelerated to minimise daily fatalities and relieve the pandemic's economic burdens, vaccine hesitancy (VH) remains a serious challenge for these efforts. VH refers to "delay in acceptance or refusal of vaccines despite availability of vaccine services",; and it is an emerging public health challenge nourished by misinformation related to vaccines effectiveness and safety. Aversion to vaccines' potential side effects is the most frequent cause of VH among population groups. Therefore, a recent systematic review revealed that raising public awareness of vaccines' effectiveness and side effects is vital for improving vaccine uptake.

Public health systems globally experience a novel and unique challenge due to the variety of vaccines manufacturers and the high levels of public awareness about those manufacturers and their marketing strategies. This unprecedented situation is predicted to create what we can refer to as "vaccine selectivity, " increasing the pressure on our weakened health systems and economies and increasing vaccine hesitancy levels. Independent (non-sponsored) studies with rigorous methods can perfectly lead the pharmacovigilance efforts of COVID-19 vaccines globally. Given their independent nature and transparent design, these studies can play a key role in suppressing vaccine hesitancy levels by enhancing public confidence in vaccines.

Design

This project comprises two phases; a) a cross-sectional survey for the short-term side effects of COVID-19 vaccines; b) a prospective cohort study for the long-term safety of COVID-19 vaccines.

Phase A:

A validated self-administered questionnaire will be developed and delivered online to the target population groups (HCW, OA & ST). The questionnaire will be inquiring about the short-term side effects that emerged within 30 days following the vaccine shot (either the first or the second dose). The side effects will be classified as local or systemic, and their onset, duration, and intensity will be self-assessed and self-reported by the respondents. This phase is proposed to take place until December 31st, 2021.

Phase B:

A validated self-administered questionnaire will be developed and delivered online to the volunteers who participated in Phase A and expressed their interest to report their long-term side effects. In this phase, the vaccine effectiveness and side effects will be evaluated after booster doses. Phase B will take place for five consecutive years starting from 2022.

ELIGIBILITY:
Inclusion Criteria:

* HCW, OA and ST who received COVID-19 vaccine.
* Participating subjects should be at least 18-year-old and able to give their informed consent independently.

Exclusion Criteria:

* Non HCW, OA and ST who received the COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In Phase A, a pragmatic approach will track each target group according to the governmental plan; in most countries, it went from HCW to OA to ST. The sample of Phase B will be pre-identified based on the outcome of Phase A. If ≥ 25% of HCW, 10% of OA and 10% of ST of Phase A showed their interest to join Phase B, no additional recruitment will be required. If < 25% of HCW, 10% of OA and 10% of ST of Phase A showed their interest in Phase B, additional recruitment will be carried out targeting healthcare workers who will receive booster doses. In case of the emergence of special side effects after booster doses, additional recruitment of healthcare workers will be required.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of local side effects (e.g. injection site pain, injection site swelling, and injection site redness)
Systemic Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of systemic side effects (e.g. fever, chills, headache, fatigue, nausea, diarrhea, etc)

SECONDARY OUTCOMES:
Unrecognized Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of oral and dermatologic side effects (e.g. oral paresthesia, oral ulcers, dysgeusia, skin rash, acne, urticaria, etc)

CONTACTS AND LOCATIONS:
Locations (14):
- American College of Physicians, Philadelphia, Pennsylvania, United States
- McMaster University, Hamilton, Ontario, Canada
- University of Split, Split, Croatia
- Masaryk University, Brno, Czechia
- University of Tartu, Tartu, Estonia
- Jimma University, Jimma, Ethiopia
- Justus-Liebig University Giessen, Giessen, Germany
- University of Ghana, Accra, Ghana
- Sinaloa's Pediatric Hospital, Culiacán, Mexico
- Medical University of Silesia, Katowice, Poland
- Nursing School of Coimbra, Coimbra, Portugal
- Irkutsk Scientific Center of Siberian Branch of Russian Academy of Sciences, Irkutsk, Russia
- University of Belgrade, Belgrade, Serbia
- University of Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riad A, Pokorna A, Attia S, Klugarova J, Koscik M, Klugar M. Prevalence of COVID-19 Vaccine Side Effects among Healthcare Workers in the Czech Republic. J Clin Med. 2021 Apr 1;10(7):1428. doi: 10.3390/jcm10071428. PMID 33916020
- [Derived] Riad A, Schunemann H, Attia S, Pericic TP, Zuljevic MF, Jurisson M, Kalda R, Lang K, Morankar S, Yesuf EA, Mekhemar M, Danso-Appiah A, Sofi-Mahmudi A, Perez-Gaxiola G, Dziedzic A, Apostolo J, Cardoso D, Marc J, Moreno-Casbas M, Wiysonge CS, Qaseem A, Gryschek A, Tadic I, Hussain S, Khan MA, Klugarova J, Pokorna A, Koscik M, Klugar M. COVID-19 Vaccines Safety Tracking (CoVaST): Protocol of a Multi-Center Prospective Cohort Study for Active Surveillance of COVID-19 Vaccines' Side Effects. Int J Environ Res Public Health. 2021 Jul 25;18(15):7859. doi: 10.3390/ijerph18157859. PMID 34360156